CLINICAL TRIAL: NCT00577018
Title: A Double-Blind, Placebo-Controlled Trial to Evaluate the Effect of Dose-Titration on the Safety and Efficacy and R108512 Tablets in Subjects With Chronic Constipation
Brief Title: Efficacy and Safety Study of the Effect of Dose-Titration of Prucalopride for The Treatment of Chronic Constipation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Movetis (Industry)
Responsible Party: Renate Specht Gryp, Movetis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRU-USA-25
Record Dates: First submitted 2007-12-17; First posted 2007-12-19 (Estimated); Last update posted 2008-05-29 (Estimated); Status verified 2007-12

CONDITIONS: Constipation
MeSH Terms: conditions — Constipation | interventions — prucalopride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator)
  Interventions: Drug: Prucalopride
- 2 (Active Comparator)
  Interventions: Drug: Prucalopride
- 3 (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Prucalopride — 4 mg o.d.
  Other Names: Resolor
  Arms: 1
Drug: Prucalopride — 1 mg o.d. for 2 days, 2 mg o.d. for 2 days and 4 mg o.d. thereafter
  Other Names: Resolor
  Arms: 2
Other: Placebo — o.d.
  Arms: 3

SUMMARY:
The purpose of this study is to determine the safety profile of 4 mg prucalopride in the treatment of chronic constipation.

DETAILED DESCRIPTION:
To evaluate the potential differences in the adverse event (safety) profile between 4 mg of prucalopride daily for 4 weeks; titration up to a 4-mg total daily dose of prucalopride by starting at 1 mg for 2 days, 2 mg for 2 days, to 4 mg thereafter; and placebo given as oral tablets once daily for 4 weeks in patients with chronic constipation

ELIGIBILITY:
Inclusion Criteria:

* Male and non-pregnant, non-breast feeding female subjects at least 18 years of age (no upper age limit);
* History of constipation. The subject reported having on average, 2 or fewer spontaneous bowel movements per week that resulted in a feeling or sensation of complete evacuation, as well as the occurrence of one or more of the following for at least 6 months before the selection visit: very hard (little balls) and/or hard stools for at least a quarter of the stools; sensation of incomplete evacuation following at least a quarter of the stools; or straining at defecation at least a quarter of the time. The above criteria only applied to spontaneous bowel movements, (i.e., not preceded within a period of 24 hours by the intake of a laxative or use of an enema). A subject who never had spontaneous bowel movements was considered to be constipated and therefore eligible for the trial;
* Constipation that was functional (i.e., not secondary to other causes);
* Willingness and ability to fill out own diary and questionnaires;
* Written informed consent, signed by the subject or legally acceptable representative and by the investigator; and
* Availability for follow-up during the trial period, as determined in the protocol.

Exclusion Criteria:

* Subjects in whom constipation was thought to be drug-induced or who were using any disallowed medication;
* Subjects suffering from secondary causes of chronic constipation. For example:

Endocrine disorders: insulin-dependent diabetes mellitus; hypopituitarism; hypothyroidism; hypercalcemia; pseudo-hypoparathyroidism; pheochromocytoma; or glucagon-producing tumors. Endocrine disorders controlled by appropriate medical therapy were not excluded, with the exception of insulin-dependent diabetes mellitus Metabolic disorders: porphyria; uremia; hypokalemia; or amyloid neuropathy. Metabolic disorders controlled by appropriate medical therapy were not excluded

• Exclusion criteria (cont'd): Neurologic disorders: Parkinson's disease; cerebral tumors; cerebrovascular accidents; multiple sclerosis; meningocele; aganglionosis; hypoganglionosis; hyperganglionosis; autonomic neuropathy; spinal cord injury; Chagas' disease; or major depression

* Presence of megacolon/megarectum or a diagnosis of pseudo-obstruction;
* Constipation as a result of surgery;
* Known or suspected organic disorders of the large bowel (i.e., obstruction, carcinoma, or inflammatory bowel disease). Results of a barium enema with flexible sigmoidoscopy or of a colonoscopic examination performed within the last 12 months were needed to rule out organic disorders. An examination performed within the last 3 years was acceptable, if the examination had been performed for an evaluation of constipation, if there was no history or evidence of weight loss, anemia, or rectal bleeding, and if the subject had had three consecutively negative stool occult blood tests at screening. Subjects with polyps discovered by colonoscopy that were untreated (i.e., by polypectomy) were to be excluded;
* Presence of severe and clinically uncontrolled cardiovascular, liver or lung disease, neurologic or psychiatric disorders (including active alcohol or drug abuse);
* Clinically significant cancer within the past 5 years;
* Known HIV-positive status or AIDS;
* Impaired renal function;
* Clinically significant abnormalities of hematology, urinalysis or blood chemistry;
* Females of child-bearing potential without adequate contraceptive protection during the trial. Oral contraceptives, Depo-Provera®, or Norplant®) must have been used for at least 3 months prior to randomization. I.U.D.'s, sterilization, or a double-barrier method were other acceptable methods of birth control;
* Treatment with an investigational drug in the 30 days preceding the run-in phase of the trial; and
* Previous treatment with either R093877 (prucalopride hydrochloride) or R108512 (prucalopride succinate).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 755 (Actual)
Dates: Start 1998-08; Primary Completion 1999-09 (Actual); Study Completion 1999-09 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with an average of ≥3 SCBM/week | 4 weeks

SECONDARY OUTCOMES:
Proportion of patients with an average increase of ≥1 SCBM/week | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: John F Johanson, MD, MSc, Principal Investigator — Private Practice